CLINICAL TRIAL: NCT02659787
Title: Effects of Buprenorphine on Mood in Adults With a Range of Depressive Symptomatology
Acronym: BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-0170
Record Dates: First submitted 2016-01-13; First posted 2016-01-20 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose buprenorphine (Active Comparator): Subjects all receive placebo, 0.2 mg buprenorphine in crossover design
  Interventions: Drug: 0.2mg Buprenorphine
- Placebo (Placebo Comparator): Subjects all receive placebo, 0.2 mg buprenorphine in crossover design
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.2mg Buprenorphine — Sublingual buprenorphine tablets (0.2mg)
  Arms: Low dose buprenorphine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study seeks to to study the effects of buprenorphine, a partial mu-opioid agonist, on depressed mood in a healthy young adults with a range of depressive symptomatology.

DETAILED DESCRIPTION:
It has been shown that opioid analgesics, particularly the mu-opioid partial agonist buprenorphine, have anti-depressant properties in laboratory animal models. In humans, rates of prescription opioid abuse are significantly higher in patients with depression. This suggests that individuals with negative mood states (e.g., depressive states) may respond more positively to opioid drugs. A handful of small studies in in humans have suggested that buprenorphine reduces symptoms of depression in patients who did not respond to standard anti-depressants, and laboratory studies have shown buprenorphine may reduce responses to some types of negative stimuli and enhance responses to positive stimuli. However, a controlled laboratory study assessing potential anti-depressant effects of an opioid medication has never been conducted. In this project, the investigators propose to examine depressive symptomatology as a predictor of subjective mood responses to buprenorphine, using two measures; i) self-reported depressive symptomatology as measured by the Beck Depression Inventory (BDI-II), and ii) physiological indices of depressive symptomatology as measured by heart rate variability. Reduced heart rate variability has been shown to be associated with depression, and such a physiological measure may allow for the detection of more subtle effects than would a self-report questionnaire alone. Healthy volunteers (N=60) will first complete the BDI and provide baseline measures of heart rate variability. Then they will attend two laboratory sessions, at which they will receive placebo or 0.2mg buprenorphine. The investigators have tested these low doses of buprenorphine in previous studies, and they produce measurable changes in mood and behavior in healthy volunteers. The investigators will collect measures of mood and physiological drug response (pupillometry, heart rate, and blood pressure) at regular intervals throughout each session, and will then examine their baseline indices of depressive symptomatology in relation to responses to the drug. The central hypothesis is that individuals with greater self-reported depressive symptoms and lower heart rate variability will experience the greatest enhancement of mood in response to buprenorphine. It is expected that this work will provide a better understanding of which individuals are most likely to experience positive mood effects in response to opioid drugs, and may therefore be at-risk for developing an opioid use disorder. Furthermore, it may lay the foundation for future research in the development of novel opioid-based treatments for depression.

Design: The study will use a 3-session within-subjects double-blind design in which participants will receive single doses of buprenorphine (0, 0.2 mg sublingual) in randomized order. All screening, orientation, and study session procedures will take place in the Human Behavioral Pharmacology Laboratory suite in the L4 wing of 5841 S. Maryland Ave.

Drug and Doses: Investigators will administer placebo, 0.2 mg buprenorphine (Temgesic) via sublingual tablet in counterbalanced order under double-blind conditions. These tablets dissolve within 5-8 minutes. This drug has been approved for treatment of severe pain. The onset of action after sublingual administration is 30 minutes, with a peak plasma concentration at 1/5-2 hours and a half-life of 5 hours. The dose of buprenorphine are very low, and the average maintenance dose for opioid abusers is 8 mg. Doses will be separated by at least 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* High school education
* Fluency in English
* BMI between 19 and 30

Exclusion Criteria:

* Medical conditions contraindicating study participation
* Regularly medication use
* Current or past opioid abuse or dependence
* Current or past drug or alcohol dependence
* Psychiatric illness
* Women who are pregnant or nursing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Falcon E, Maier K, Robinson SA, Hill-Smith TE, Lucki I. Effects of buprenorphine on behavioral tests for antidepressant and anxiolytic drugs in mice. Psychopharmacology (Berl). 2015 Mar;232(5):907-15. doi: 10.1007/s00213-014-3723-y. Epub 2014 Sep 3. PMID 25178815
- [Background] Sullivan MD, Edlund MJ, Steffick D, Unutzer J. Regular use of prescribed opioids: association with common psychiatric disorders. Pain. 2005 Dec 15;119(1-3):95-103. doi: 10.1016/j.pain.2005.09.020. Epub 2005 Nov 17. PMID 16298066
- [Background] Karp JF, Butters MA, Begley AE, Miller MD, Lenze EJ, Blumberger DM, Mulsant BH, Reynolds CF 3rd. Safety, tolerability, and clinical effect of low-dose buprenorphine for treatment-resistant depression in midlife and older adults. J Clin Psychiatry. 2014 Aug;75(8):e785-93. doi: 10.4088/JCP.13m08725. PMID 25191915
- [Background] Nyhuis PW, Gastpar M, Scherbaum N. Opiate treatment in depression refractory to antidepressants and electroconvulsive therapy. J Clin Psychopharmacol. 2008 Oct;28(5):593-5. doi: 10.1097/JCP.0b013e31818638a4. No abstract available. PMID 18794671
- [Background] Bodkin JA, Zornberg GL, Lukas SE, Cole JO. Buprenorphine treatment of refractory depression. J Clin Psychopharmacol. 1995 Feb;15(1):49-57. doi: 10.1097/00004714-199502000-00008. PMID 7714228
- [Background] Striebel JM, Kalapatapu RK. The anti-suicidal potential of buprenorphine: a case report. Int J Psychiatry Med. 2014;47(2):169-74. doi: 10.2190/PM.47.2.g. PMID 25084802
- [Background] Licht CM, de Geus EJ, Zitman FG, Hoogendijk WJ, van Dyck R, Penninx BW. Association between major depressive disorder and heart rate variability in the Netherlands Study of Depression and Anxiety (NESDA). Arch Gen Psychiatry. 2008 Dec;65(12):1358-67. doi: 10.1001/archpsyc.65.12.1358. PMID 19047522
- [Background] Ipser JC, Terburg D, Syal S, Phillips N, Solms M, Panksepp J, Malcolm-Smith S, Thomas K, Stein DJ, van Honk J. Reduced fear-recognition sensitivity following acute buprenorphine administration in healthy volunteers. Psychoneuroendocrinology. 2013 Jan;38(1):166-70. doi: 10.1016/j.psyneuen.2012.05.002. Epub 2012 May 30. PMID 22651957

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Buprenorphine: Participants first received placebo during first study session. After a washout period of 3 days, participants returned to lab and they then received 0.2 mg buprenorphine (Sublingual buprenorphine tablets (0.2mg).
- Buprenorphine, Then Placebo: Participants first received 0.2 mg buprenorphine (Sublingual buprenorphine tablets (0.2mg) during first study session. After a washout period of 3 days, participants returned to lab and they received placebo tablet.
Period: First Intervention (1 Day)
Arm/Group | Placebo, Then Buprenorphine | Buprenorphine, Then Placebo
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Washout (3 Days)
Arm/Group | Placebo, Then Buprenorphine | Buprenorphine, Then Placebo
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo, Then Buprenorphine | Buprenorphine, Then Placebo
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ALL Subjects: Subjects all receive placebo, 0.2 mg buprenorphine in crossover design
Arm/Group | ALL Subjects
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 20
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Subscales of the Drug Effects Questionnaire Subjective Response With and Without Buprenorphine
Description: The Drug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", and "Want More". The "Feel Drug", "Feel High", "Like Drug", and "Want More" subscales are reported. All subscales are scored on a visual analogue scale (scroll bar on computer screen) ranging from 0 -100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: 0 through 3 hours after dosing.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low Dose Buprenorphine | Placebo
Number analyzed (Participants) | 38 | 38
units on a scale
  Feel Drug | 21.03 (3.32) | 10.64 (2.42)
  Like Drug | 23.09 (3.97) | 19.8 (4.12)
  Feel High | 10.91 (2.44) | 5.74 (1.62)
  Want More | 17.46 (3.90) | 16.76 (3.86)

ADVERSE EVENTS:
Time Frame: 6 days for each intervention
Groups:
- Placebo, Then Buprenorphine: Participants first received placebo during first study session. After a washout period of 3 days, participants returned to lab and they then received 0.2 mg buprenorphine (sublingual buprenorphine tablets (0.2 mg).
- Buprenorphine, Then Placebo: Participants first received 0.2 mg buprenorphine (Sublingual buprenorphine tablets (0.2 mg)) during first study session. After a washout period of 3 days, participants returned to lab and they then received placebo tablet.
Arm/Group | Placebo, Then Buprenorphine | Buprenorphine, Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT02659787/Prot_SAP_000.pdf